CLINICAL TRIAL: NCT04210232
Title: Post-market Evaluation of Surgeon Feedback on TECNIS® TORIC II Intraocular Lens (IOL)
Brief Title: Post-market Study to Obtain Surgeon Feedback on Clinical Outcome in Eyes Implanted With TECNIS Toric II IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NXGT-201-TTL2
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TECNIS® TORIC II Intraocular Lens (IOL) (Experimental): Subjects will be implanted with the TECNIS Toric II IOL in one or both eyes qualified for study inclusion
  Interventions: Device: TECNIS® TORIC II Intraocular Lens (IOL)

INTERVENTIONS:
Device: TECNIS® TORIC II Intraocular Lens (IOL) — Surgeons will perform standardized, small-incision, cataract surgery and implant in one or both eyes the study lenses.

SUMMARY:
This is a multicenter, prospective, single-arm, open-label, clinical study of the commercially available TECNIS Toric II, Model ZCU IOL. The study will be conducted in up to 1100 subjects enrolled with 1,000 subjects needing unilateral or bilateral cataract surgery across up to 50 US study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or bilateral cataracts for which phacoemulsification extraction and posterior chamber IOL implantation have been planned;
2. Preoperative corneal astigmatism of one diopter or more in the operative eye;
3. Potential for postoperative best corrected distance visual acuity (BCDVA) of 20/30 Snellen or better;
4. Clear intraocular media other than cataract in each eye;
5. Ability to understand, read and write English in order to consent to study participation;
6. Availability, willingness, sufficient cognitive awareness to comply with examination procedures;
7. Signed Informed Consent Document (ICD) and Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

1. Recurrent severe anterior or posterior segment inflammation or uveitis;
2. Compromised eye due to previous trauma or developmental defects in which appropriate support of the IOL is not possible;
3. Circumstances that would result in damage to the endothelium during implantation;
4. Suspected ocular microbial infection;
5. Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects;
6. Known ocular disease or pathology that, in the opinion of the investigator, may affect visual acuity or require surgical intervention during the course of the study, [macular degeneration, cystoid macular edema, proliferative diabetic retinopathy (severe), uncontrolled glaucoma, irregular corneal astigmatism, choroidal hemorrhage, concomitant severe eye disease, extremely shallow anterior chamber, microphthalmos, non-age related cataract, severe corneal dystrophy, severe optic nerve atrophy, etc.];
7. Planned monovision correction;
8. Concurrent participation or participation within 30 days prior to the preoperative visit in any other clinical study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (12):
- United States (12):
  - Empire Eye & Laser Center, Bakersfield, California
  - Jones Eye Clinic, Sioux City, Iowa
  - Chesapeake Eye Care and Laser Center, Annapolis, Maryland
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Oakland Ophthalmic Surgery, P.C., Birmingham, Michigan
  - Tekwani Vision Center, St Louis, Missouri
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Key & Whitman Eye Center, Dallas, Texas
  - Texas Eye and Laser Center, Hurst, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Clarus Eye Center, Lacey, Washington

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 87 subjects signed informed consent in the study. 33 were screen failures and 54 subjects were treated/implanted across 8 clinical sites in the US. Of the 54 subjects treated, 32 subjects were treated bilaterally, and 22 subjects were treated unilaterally.
Groups:
- TECNIS Toric II: Study Lens
Period: Overall Study
Arm/Group | TECNIS Toric II
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TECNIS Toric II
Number analyzed (Participants) | 54
Age, Customized [Number; unit: Participants]
  <60 years | 3
  60-69 years | 19
  70-79 years | 25
  >=80 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1
  African American | 2
  Native hawaiian/Pacific islander | 0
  Caucasian | 51
  Other | 0
  Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Surgeon Satisfaction of the Clinical Outcome of Eye Implanted With the TECNIS Toric II
Description: Percent of Eyes Rated Very Satisfied or Satisfied with Clinical Outcomes. This endpoint was assessed based on the question "Please rate your overall level of satisfaction with the clinical outcomes achieved in the implanted eye" in the Surgeon Satisfaction Questionnaire (SSQ).
Time Frame: 3 months postoperative
Population: All Toric II Eyes
Measure: Number (95% Confidence Interval); unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | TECNIS Toric II
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 85
Percentage of eyes
  Very Satisfied/Satisfied | 100 [95.8 to 100]
  Undecided/Dissatisfied/Very Dissatisfied | 0 [0 to 4.2]

ADVERSE EVENTS:
Time Frame: 3 months postoperative
Arm/Group | TECNIS Toric II
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 6/54
Other Adverse Events (participants affected / at risk) | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TECNIS Toric II (N=54)
Hospitalization due to bleeding varices (Gastrointestinal disorders) | 1 (1)
Hospitalization due to heart attack (Cardiac disorders) | 2 (2)
Cystoid Macular Edema (Eye disorders) | 1 (1)
Hospitalization (Renal and urinary disorders) | 1 (1)
Hospitalization due to vomiting of blood (Gastrointestinal disorders) | 1 (1)
Hospitalization due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04210232/Prot_SAP_000.pdf